CLINICAL TRIAL: NCT03017534
Title: Non-Specific Effects of Manual Therapy: A Mixed-Methods Investigation of Contextual and Social Interactions
Brief Title: Non-Specific Effects of Manual Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shenandoah University (Other)
Responsible Party: Principal Investigator, Aaron Hartstein, Assistant Professor, Division of Physical Therapy, Shenandoah University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ShenandoahU (2)
Record Dates: First submitted 2017-01-09; First posted 2017-01-11 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Musculoskeletal Manipulations; Placebo Effect
Keywords: Patient-Therapist Interaction; Non-Specific Effects; Manual Therapy; Neurodynamics; Sham

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (8):
- Gender Match, Labcoat, Explanation (Experimental): Subjects will receive Spinal Manual Therapy (sham thoracic spine manipulation) by a gender matched therapist, wearing a labcoat and receive a detailed anatomic explanation of the technique.
  Interventions: Procedure: Spinal Manual Therapy
- Gender Match, Labcoat, No Explanation (Experimental): Subjects will receive Spinal Manual Therapy (sham thoracic spine manipulation) by a gender matched therapist, wearing a labcoat, and receive a colloquial discussion of the technique.
  Interventions: Procedure: Spinal Manual Therapy
- Gender Match, No Labcoat, Explanation (Experimental): Subjects will receive Spinal Manual Therapy (sham thoracic spine manipulation) by a gender matched therapist, not wearing a labcoat, and receive a detailed anatomic explanation of the technique.
  Interventions: Procedure: Spinal Manual Therapy
- Gender Match, No Labcoat, No Explanation (Experimental): Subjects will receive Spinal Manual Therapy (sham thoracic spine manipulation) by a gender matched therapist, not wearing a labcoat, and receive a colloquial discussion of the technique.
  Interventions: Procedure: Spinal Manual Therapy
- Gender Mis-match, Labcoat, Explanation (Experimental): Subjects will receive Spinal Manual Therapy (sham thoracic spine manipulation) by a gender mis-matched therapist, wearing a labcoat and receive a detailed anatomic explanation of the technique.
  Interventions: Procedure: Spinal Manual Therapy
- Gender Mis-match, Labcoat, No Explan. (Experimental): Subjects will receive Spinal Manual Therapy (sham thoracic spine manipulation) by a gender mis-matched therapist, wearing a labcoat, and receive a colloquial discussion of the technique.
  Interventions: Procedure: Spinal Manual Therapy
- Gender Mis-match, No Labcoat, Explan. (Experimental): Subjects will receive Spinal Manual Therapy (sham thoracic spine manipulation) by a gender mis-matched therapist, not wearing a labcoat, and receive a detailed anatomic explanation of the technique.
  Interventions: Procedure: Spinal Manual Therapy
- Gender Mis-match, No Labcoat, No Explan. (Experimental): Subjects will receive Spinal Manual Therapy (sham thoracic spine manipulation) by a gender matched therapist, not wearing a labcoat, and receive a colloquial discussion of the technique.
  Interventions: Procedure: Spinal Manual Therapy

INTERVENTIONS:
Procedure: Spinal Manual Therapy — Supine thoracic spine sham manipulation located between the levels of T4-7; identical procedure as an active treatment intervention but without the delivery of a high velocity low amplitude thrust

SUMMARY:
The mechanism responsible for improvement following manual physical therapy techniques is unknown. Previous studies have indicated both biomechanical and neurophysiologic effects which may be responsible for clinical changes observed. Yet, other studies report clinical changes following sham interventions. Through a mixed-methods design, this study aims to gain more understanding of the social and contextual factors that may be related to the improvement often observed following manual therapy techniques.

DETAILED DESCRIPTION:
A convenience sample will be utilized to obtain subjects. Subjects will be given a brief questionnaire to identify possible contraindications for manual therapy treatment techniques and exclude individuals if necessary. Subjects will be randomized into one of eight groups (three variables, each with two conditions including: therapist gender match/mismatch, lab coat worn/not worn, detailed explanation/colloquial conversation about the technique) and participate in neurodynamic testing for the upper quarter via the Upper Limb Provocation Test. Subjects who are determined to be positive for one or more extremities will receive a sham thoracic spine manipulation technique. After application of the technique, previously positive limbs will be retested. Individuals who respond favorably to the sham technique upon reassessment will participate in an exit interview with open-ended questions in attempt to gain more insight into the factors which may have influenced their neurodynamic mobility improvement.

ELIGIBILITY:
Inclusion Criteria:

* Upper Limb Provocation Test results with limitation greater than 60 deg of elbow extension at the time of measurement

Exclusion Criteria:

* History of cervical or lumbar pain requiring medical intervention within the last two years, history of upper or lower extremity paresthesia/numbness, self reported bone density disorders, previous spinal cord injury, diagnosed intervertebral disc herniation, previous diagnosis of spinal stenosis or disc pathology, current pregnancy, history of circulatory or neurological disorders, history of spine and extremity fractures or dislocations in the last two years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Change in Upper Limb Provocation Test (ULPT) | Baseline and Immediately Post Intervention
  Subjects will lie on their back with their shoulder slightly off the edge of a treatment table. The investigator will sidebend the subjects neck away from the extremity being tested and gradually move the extremity into the following positions: scapular depression, shoulder 90 deg abduction, shoulder 90 deg external rotation, forearm supination, wrist/finger extension, and elbow extension. The investigator will assess for symptoms at each phase throughout the test. At the onset of symptoms, sensitization maneuvers will be completed to determine if the origin of the symptoms is neurodynamic in nature and not myofascial.

CONTACTS AND LOCATIONS:
Overall Officials: Sheri A Hale, PT, PhD, ATC, Study Director — Shenandoah University
Locations (1):
- Shenandoah University, Winchester, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bialosky JE, Bishop MD, George SZ, Robinson ME. Placebo response to manual therapy: something out of nothing? J Man Manip Ther. 2011 Feb;19(1):11-9. doi: 10.1179/2042618610Y.0000000001. PMID 22294849
- [Background] Bialosky JE, Bishop MD, Price DD, Robinson ME, George SZ. The mechanisms of manual therapy in the treatment of musculoskeletal pain: a comprehensive model. Man Ther. 2009 Oct;14(5):531-8. doi: 10.1016/j.math.2008.09.001. Epub 2008 Nov 21. PMID 19027342
- [Background] O'Keeffe M, Cullinane P, Hurley J, Leahy I, Bunzli S, O'Sullivan PB, O'Sullivan K. What Influences Patient-Therapist Interactions in Musculoskeletal Physical Therapy? Qualitative Systematic Review and Meta-Synthesis. Phys Ther. 2016 May;96(5):609-22. doi: 10.2522/ptj.20150240. Epub 2015 Oct 1. PMID 26427530
- [Background] Testa M, Rossettini G. Enhance placebo, avoid nocebo: How contextual factors affect physiotherapy outcomes. Man Ther. 2016 Aug;24:65-74. doi: 10.1016/j.math.2016.04.006. Epub 2016 Apr 20. PMID 27133031
- [Result] Davis DS, Anderson IB, Carson MG, Elkins CL, Stuckey LB. Upper Limb Neural Tension and Seated Slump Tests: The False Positive Rate among Healthy Young Adults without Cervical or Lumbar Symptoms. J Man Manip Ther. 2008;16(3):136-41. doi: 10.1179/jmt.2008.16.3.136. PMID 19119402